CLINICAL TRIAL: NCT02137928
Title: Carboplatin Periocular Injection in the Treatment for Retinoblastoma--A Single Center, Randomized Study to Evaluate the Efficacy of Carboplatin in Subjects With Retinoblastoma
Brief Title: Carboplatin Periocular Injection for Retinoblastoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yanghs2014
Record Dates: First submitted 2014-05-10; First posted 2014-05-14 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-08

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; carboplatin
MeSH Terms: conditions — Retinoblastoma | interventions — Carboplatin; Vincristine; Etoposide; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carboplatin periocular injection (Experimental): 20mg/2ml carboplatin periocular injection together with CEV chemotherapy(CEV Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months)
  Interventions: Drug: carboplatin periocular injection
- chemotherapy (Active Comparator): Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: carboplatin periocular injection — 20mg/2ml carboplatin periocular injection together with chemotherapy
  Other Names: carboplatin; vincristine, carboplatin, etoposide
  Arms: carboplatin periocular injection
Drug: chemotherapy — Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months.
  Other Names: vincristine, carboplatin, etoposide
  Arms: chemotherapy

SUMMARY:
This study will evaluate the clinical efficacy of periocular injections of carboplatin together with chemotherapy in the treatment of Retinoblastoma as compared to chemotherapy alone.

DETAILED DESCRIPTION:
This study will be a phase Ⅲ open label interventional case series. Patients with retinoblastoma will be randomized to receive chemotherapy with or without periocular injections of carboplatin at a dose of 20mg/2 ml. Patients will receive carboplatin periocular on a monthly basis for a total duration of therapy of 6 months. Patients will be followed for 24 months .

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* linical diagnosis of retinoblastoma, Stage 0 or Ⅱ base on International Retinoblastoma Staging System.

Exclusion Criteria:

* Any previous disease in the study eye.
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals).
* History of chemical intervention for retinoblastoma in the study eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | two years
  measure the mortality rate for the two groups(Cancer-related death and non-Cancer-related death) at two years

SECONDARY OUTCOMES:
side effects of carboplatin periocular injection in the Treatment of Retinoblastoma | two years
  Measure the side effects(systemic check-up, local side effects) before each treatment, and 1,3,6,9,12,18,24 months after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, Doctor, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China